CLINICAL TRIAL: NCT00469391
Title: A Multi-Center, Pilot Efficacy Study of the GI Sleeve for Pre-Surgical Weight Loss
Brief Title: Multi-Center Pre-Bariatric Weight Loss Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-3
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Results first posted 2016-12-30 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Obesity
Keywords: Weight Reduction
MeSH Terms: conditions — Obesity; Weight Loss | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GI Sleeve (Experimental): medical device that mimics gastric bypass mechanism for weight-loss
  Interventions: Device: GI Sleeve Implantable weight loss device (EndoBarrier)
- Sham Control (Sham Comparator)
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Device: GI Sleeve Implantable weight loss device (EndoBarrier) — device for weight loss
  Other Names: endobarrier
  Arms: GI Sleeve
Procedure: Sham Procedure — Weight loss
  Other Names: Sham
  Arms: Sham Control

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of the GI Sleeve in patients who require weight loss prior to their Bariatric surgery.

DETAILED DESCRIPTION:
This is a randomized, patient blinded, prospective study.Patients will receive either a device or a sham procedure. Patients will be evaluated for the study and randomized to a treatment group if they qualify for the study. Throughout the study their weights will be obtained and various laboratory tests collected. A comparison of weight loss between the two groups will be assessed as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35 with a significant comorbid condition or BMI 40-60
* Candidate for Bariatric Surgery

Exclusion Criteria:

* No pathologies of the GI Tract
* No anti-coagulant or non-steroidal anti-inflammatory medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tarnoff, MD, Study Director — Tufts Medical Center
Locations (4):
- United States (4):
  - Cleveland Clinic Florida, Weston, Florida
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Carolinas Medical Center, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual patient data is on file at the Sponsor

RESULTS

PARTICIPANT FLOW:
Groups:
- GI Sleeve: GI Sleeve Implantable weight loss device (EndoBarrier): device for weight loss followed by standard-of-care diet therapy
- Sham Control: Sham Procedure followed by standard-of-care diet therapy
Period: Overall Study
Arm/Group | GI Sleeve | Sham Control
Started | 27 | 29
Discontinued Prior to Procedure | 2 | 3
Unsuccessful Implant Procedure | 4 | 0
Adverse Event | 8 | 0
Lost to Follow up | 0 | 1
Patient Preference | 0 | 1
Completed | 13 | 24
Not Completed | 14 | 5

BASELINE CHARACTERISTICS:
Population: ITT population: All subjects who did not withdraw before the procedure and device subjects who had a successful implant procedure
Groups:
- Total: Total of all reporting groups
Arm/Group | GI Sleeve | Sham Control | Total
Number analyzed (Participants) | 21 | 26 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (7.4) | 42.7 (9.5) | 43.7 (8.8)
Gender [Count of Participants; unit: Participants]
  Female | 15 | 23 | 38
  Male | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 21 | 26 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percent Excess Weight Loss (%EWL) at Week 12
Description: Excess Weight Loss was calculated using the Metropolitan Life Table (MET method)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Percentage of Excess Weight Loss
Arm/Group | GI Sleeve | Sham Control
Number analyzed (Participants) | 13 | 24
Percentage of Excess Weight Loss | 11.9 (1.4) | 2.7 (2.0)

ADVERSE EVENTS:
Groups:
- GI Sleeve: N=26 for attempted device implant procedures. There were 2 subjects who withdrew from the study before the procedure and 4 unsuccessful procedure. Thus, N=21 for ITT population ( subjects with implanted devices).
- Sham Control: 3 subjects withdrew before the procedure. N=26 for the ITT population.
Arm/Group | GI Sleeve | Sham Control
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/26
Other Adverse Events (participants affected / at risk) | 21/21 | 20/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GI Sleeve (N=21) | Sham Control (N=26)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GI Sleeve (N=21) | Sham Control (N=26)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 9 (9) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6) | 5 (5)
Adverse drug reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pharyngolaryngeal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Procedural Nausea (Injury, poisoning and procedural complications) | 16 (16) | 6 (6)
Procedural vomiting (Injury, poisoning and procedural complications) | 7 (7) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Upper Respiratory Tract infection (Infections and infestations) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No